CLINICAL TRIAL: NCT01049867
Title: Phase 1-2 Study of Intracoronary Infusion of CD133+ Endothelial Precursor Cells for Patients With Coronary Heart Disease in Selected Obstructed Artery
Brief Title: CD133+ Cell Therapy for Refractory Coronary Heart Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital y Clinica OCA, S.A. de C.V. (Other)
Responsible Party: Dr. Genaro Levinson/Director, Hospital y Clinica OCA, S.A. de C.V.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASOR01CMN093300CT051044-1895; CASOR01CMN093300CT051044-1895 (Other: COFEPRIS, Mexican Secretariat of Health)
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intracoronary Infusion of CD133+ Cells — Single intracoronary infusion of a suspension consisting of 30 ml saline solution containing at least 1 million CD133+ endothelial precursor cells.

SUMMARY:
The aim of this study is to evaluate if the intracoronary infusion of autologous bone-marrow derived CD133+ endothelial precursor cells is able to promote neovascularization and to improve myocardial perfusion and contractility in patients with refractory coronary heart disease, characterized by poor response to standard coronary interventions, severe impairment of the quality of life, and poor prognosis.

DETAILED DESCRIPTION:
Refractory Coronary Artery Disease is a significant cause of mortality and decreased quality of life. Intracoronary infusion of CD133+ progenitor cells is a viable treatment option for patients with this condition. After clinical and laboratory evaluation, 50-100 ml of bone marrow will be obtained by bone marrow aspiration from the posterior iliac crest under local anesthesia. From this sample, CD133+ endothelial progenitor cells will be isolated, purified and packed within the next 12 hours of extraction, and resuspended in 30 ml saline solution. The patient will undergo coronary catheterization for selection of the target obstructed artery for cell infusion, which will be performed using a balloon catheter under hemodynamic monitoring. Once concluded, the patient will be transferred to intermediate care unit for post-interventional observation for approximately 24 hours before being released. Ambulatory follow-up will be performed at specific intervals to determine efficacy and safety of this intervention by clinical and laboratory examination, including imaging and cardiac function studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven CHD by coronary angiography demonstrating occlusion or extreme stenosis (> 90%) of a coronary artery (target artery) not suitable for angioplasty or surgery.
* Angiographic criteria: Feasibility for balloon catheter placement without risks of obstruction of the left main coronary trunk.
* Evidence of viable myocardial tissue in the area irrigated by the target artery by MRI (low dose dobutamine and late enhancement).
* CCS class 2-4 angina pectoris (angina pectoris at rest and at light exertion, obvious reduction in the exertion capacity).
* Optimal antianginal pharmacologic therapy (consistent with the current guidelines of ACC (American College of Cardiology), as well as the DGK (Deutsche Gesellschaft für Kardiologie)
* Signed written consent form accepted by the Ethics Committee.
* Effective contraception in women of child-bearing age.

Exclusion Criteria:

* Severe symptomatic heart failure (NYHA class 4).
* Myocardial aneurysm (in the target region) without evidence of viable myocardium.
* Myocardial infarction in the last 4 weeks.
* Symptomatic ventricular tachycardia.
* Known malignancy.
* Known hematological disease.
* Renal insufficiency with creatinine > 2.5 mg/dl.
* Pregnancy.
* Active chronic inflammatory bowel disease or rheumatic disease with high parameters of inflammation (WBCs above 10/nl and increased C-reactive protein). Systemic steroid administration.
* Severe coagulopathy or phenprocoumon type anticoagulation therapy at the time of bone marrow extraction.
* Antiproliferative therapy (chemotherapy, etc.).
* Non accordance with procedures and follow-up studies.
* Contraindications to MRI studies.
* Known hypersensitivity against mouse immunoglobulins.
* Known hypersensitivity against ferridextran.
* Contraindications for bone marrow extraction.
* Cerebrovascular accident in the past four months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Increased regional and global myocardial contractility measured by low-dose dobutamine echocardiography/MRI and increased myocardial perfusion measured by adenosine nuclear stress testing. | Base-line, 3, and 6 months.

SECONDARY OUTCOMES:
Improvement in the heart failure functional class measured by NYHA and CCS classification tests. | Base-line, 3, and 6 months
Changes in the score of the "Minnessota living with heart failure score". | Base-line, 3, and 6 months.
Functional heart changes measured by spiroergometry. | Base-line, 3, and 6 months.
Reduction in the consumption of medicines for the heart ailment (nitrates, diuretics, etc.). | Base-line, 3, and 6 months.
Safety and compatibility through evaluation of adverse events (death, supraventricular and ventricular arrhythmias, brain/peripheral ischemic events, myocardial infarct, malignancies, etc.). | Base-line, 3, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Rojas-Martinez, M.D./D.Sc., Study Chair — Director, Cell Therapy Laboratory. OCA Hospital
Locations (1):
- Hospital y Clinica OCA, S.A de C.V., Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Pittenger MF, Mackay AM, Beck SC, Jaiswal RK, Douglas R, Mosca JD, Moorman MA, Simonetti DW, Craig S, Marshak DR. Multilineage potential of adult human mesenchymal stem cells. Science. 1999 Apr 2;284(5411):143-7. doi: 10.1126/science.284.5411.143. PMID 10102814
- [Background] Krause DS, Theise ND, Collector MI, Henegariu O, Hwang S, Gardner R, Neutzel S, Sharkis SJ. Multi-organ, multi-lineage engraftment by a single bone marrow-derived stem cell. Cell. 2001 May 4;105(3):369-77. doi: 10.1016/s0092-8674(01)00328-2. PMID 11348593
- [Background] Jackson KA, Majka SM, Wang H, Pocius J, Hartley CJ, Majesky MW, Entman ML, Michael LH, Hirschi KK, Goodell MA. Regeneration of ischemic cardiac muscle and vascular endothelium by adult stem cells. J Clin Invest. 2001 Jun;107(11):1395-402. doi: 10.1172/JCI12150. PMID 11390421
- [Background] Jiang Y, Jahagirdar BN, Reinhardt RL, Schwartz RE, Keene CD, Ortiz-Gonzalez XR, Reyes M, Lenvik T, Lund T, Blackstad M, Du J, Aldrich S, Lisberg A, Low WC, Largaespada DA, Verfaillie CM. Pluripotency of mesenchymal stem cells derived from adult marrow. Nature. 2002 Jul 4;418(6893):41-9. doi: 10.1038/nature00870. Epub 2002 Jun 20. PMID 12077603
- [Background] Orlic D, Kajstura J, Chimenti S, Bodine DM, Leri A, Anversa P. Transplanted adult bone marrow cells repair myocardial infarcts in mice. Ann N Y Acad Sci. 2001 Jun;938:221-9; discussion 229-30. doi: 10.1111/j.1749-6632.2001.tb03592.x. PMID 11458511
- [Background] Wang JS, Shum-Tim D, Chedrawy E, Chiu RC. The coronary delivery of marrow stromal cells for myocardial regeneration: pathophysiologic and therapeutic implications. J Thorac Cardiovasc Surg. 2001 Oct;122(4):699-705. doi: 10.1067/mtc.2001.116317. PMID 11581601
- [Background] Orlic D, Kajstura J, Chimenti S, Bodine DM, Leri A, Anversa P. Bone marrow stem cells regenerate infarcted myocardium. Pediatr Transplant. 2003;7 Suppl 3:86-8. doi: 10.1034/j.1399-3046.7.s3.13.x. PMID 12603699
- [Background] Orlic D, Kajstura J, Chimenti S, Jakoniuk I, Anderson SM, Li B, Pickel J, McKay R, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Bone marrow cells regenerate infarcted myocardium. Nature. 2001 Apr 5;410(6829):701-5. doi: 10.1038/35070587. PMID 11287958
- [Background] Orlic D, Kajstura J, Chimenti S, Limana F, Jakoniuk I, Quaini F, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Mobilized bone marrow cells repair the infarcted heart, improving function and survival. Proc Natl Acad Sci U S A. 2001 Aug 28;98(18):10344-9. doi: 10.1073/pnas.181177898. Epub 2001 Aug 14. PMID 11504914
- [Background] Wollert KC, Drexler H. Clinical applications of stem cells for the heart. Circ Res. 2005 Feb 4;96(2):151-63. doi: 10.1161/01.RES.0000155333.69009.63. PMID 15692093
- [Background] Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Assmus B, Tonn T, Dimmeler S, Zeiher AM; REPAIR-AMI Investigators. Intracoronary bone marrow-derived progenitor cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1210-21. doi: 10.1056/NEJMoa060186. PMID 16990384
- [Background] Assmus B, Schachinger V, Teupe C, Britten M, Lehmann R, Dobert N, Grunwald F, Aicher A, Urbich C, Martin H, Hoelzer D, Dimmeler S, Zeiher AM. Transplantation of Progenitor Cells and Regeneration Enhancement in Acute Myocardial Infarction (TOPCARE-AMI). Circulation. 2002 Dec 10;106(24):3009-17. doi: 10.1161/01.cir.0000043246.74879.cd. PMID 12473544
- [Background] Drexler H, Meyer GP, Wollert KC. Bone-marrow-derived cell transfer after ST-elevation myocardial infarction: lessons from the BOOST trial. Nat Clin Pract Cardiovasc Med. 2006 Mar;3 Suppl 1:S65-8. doi: 10.1038/ncpcardio0407. PMID 16501634
- [Background] Meyer GP, Wollert KC, Lotz J, Steffens J, Lippolt P, Fichtner S, Hecker H, Schaefer A, Arseniev L, Hertenstein B, Ganser A, Drexler H. Intracoronary bone marrow cell transfer after myocardial infarction: eighteen months' follow-up data from the randomized, controlled BOOST (BOne marrOw transfer to enhance ST-elevation infarct regeneration) trial. Circulation. 2006 Mar 14;113(10):1287-94. doi: 10.1161/CIRCULATIONAHA.105.575118. Epub 2006 Mar 6. PMID 16520413
- [Background] Schaefer A, Meyer GP, Fuchs M, Klein G, Kaplan M, Wollert KC, Drexler H. Impact of intracoronary bone marrow cell transfer on diastolic function in patients after acute myocardial infarction: results from the BOOST trial. Eur Heart J. 2006 Apr;27(8):929-35. doi: 10.1093/eurheartj/ehi817. Epub 2006 Mar 1. PMID 16510465
- [Background] Wollert KC, Meyer GP, Lotz J, Ringes-Lichtenberg S, Lippolt P, Breidenbach C, Fichtner S, Korte T, Hornig B, Messinger D, Arseniev L, Hertenstein B, Ganser A, Drexler H. Intracoronary autologous bone-marrow cell transfer after myocardial infarction: the BOOST randomised controlled clinical trial. Lancet. 2004 Jul 10-16;364(9429):141-8. doi: 10.1016/S0140-6736(04)16626-9. PMID 15246726
- [Background] Janssens S, Dubois C, Bogaert J, Theunissen K, Deroose C, Desmet W, Kalantzi M, Herbots L, Sinnaeve P, Dens J, Maertens J, Rademakers F, Dymarkowski S, Gheysens O, Van Cleemput J, Bormans G, Nuyts J, Belmans A, Mortelmans L, Boogaerts M, Van de Werf F. Autologous bone marrow-derived stem-cell transfer in patients with ST-segment elevation myocardial infarction: double-blind, randomised controlled trial. Lancet. 2006 Jan 14;367(9505):113-21. doi: 10.1016/S0140-6736(05)67861-0. PMID 16413875
- [Background] Fernandez-Aviles F, San Roman JA, Garcia-Frade J, Fernandez ME, Penarrubia MJ, de la Fuente L, Gomez-Bueno M, Cantalapiedra A, Fernandez J, Gutierrez O, Sanchez PL, Hernandez C, Sanz R, Garcia-Sancho J, Sanchez A. Experimental and clinical regenerative capability of human bone marrow cells after myocardial infarction. Circ Res. 2004 Oct 1;95(7):742-8. doi: 10.1161/01.RES.0000144798.54040.ed. Epub 2004 Sep 9. PMID 15358665
- [Background] Chen SL, Fang WW, Ye F, Liu YH, Qian J, Shan SJ, Zhang JJ, Chunhua RZ, Liao LM, Lin S, Sun JP. Effect on left ventricular function of intracoronary transplantation of autologous bone marrow mesenchymal stem cell in patients with acute myocardial infarction. Am J Cardiol. 2004 Jul 1;94(1):92-5. doi: 10.1016/j.amjcard.2004.03.034. PMID 15219514
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Perin EC, Dohmann HF, Borojevic R, Silva SA, Sousa AL, Mesquita CT, Rossi MI, Carvalho AC, Dutra HS, Dohmann HJ, Silva GV, Belem L, Vivacqua R, Rangel FO, Esporcatte R, Geng YJ, Vaughn WK, Assad JA, Mesquita ET, Willerson JT. Transendocardial, autologous bone marrow cell transplantation for severe, chronic ischemic heart failure. Circulation. 2003 May 13;107(18):2294-302. doi: 10.1161/01.CIR.0000070596.30552.8B. Epub 2003 Apr 21. PMID 12707230
- [Background] Patel AN, Geffner L, Vina RF, Saslavsky J, Urschel HC Jr, Kormos R, Benetti F. Surgical treatment for congestive heart failure with autologous adult stem cell transplantation: a prospective randomized study. J Thorac Cardiovasc Surg. 2005 Dec;130(6):1631-8. doi: 10.1016/j.jtcvs.2005.07.056. Epub 2005 Oct 26. PMID 16308009
- [Background] Rafii S, Lyden D. Therapeutic stem and progenitor cell transplantation for organ vascularization and regeneration. Nat Med. 2003 Jun;9(6):702-12. doi: 10.1038/nm0603-702. PMID 12778169
- [Background] Stamm C, Westphal B, Kleine HD, Petzsch M, Kittner C, Klinge H, Schumichen C, Nienaber CA, Freund M, Steinhoff G. Autologous bone-marrow stem-cell transplantation for myocardial regeneration. Lancet. 2003 Jan 4;361(9351):45-6. doi: 10.1016/S0140-6736(03)12110-1. PMID 12517467
- [Background] Klein HM, Ghodsizad A, Marktanner R, Poll L, Voelkel T, Mohammad Hasani MR, Piechaczek C, Feifel N, Stockschlaeder M, Burchardt ER, Kar BJ, Gregoric I, Gams E. Intramyocardial implantation of CD133+ stem cells improved cardiac function without bypass surgery. Heart Surg Forum. 2007;10(1):E66-9. doi: 10.1532/HSF98.20061054. PMID 17162408
- [Background] Bartunek J, Vanderheyden M, Vandekerckhove B, Mansour S, De Bruyne B, De Bondt P, Van Haute I, Lootens N, Heyndrickx G, Wijns W. Intracoronary injection of CD133-positive enriched bone marrow progenitor cells promotes cardiac recovery after recent myocardial infarction: feasibility and safety. Circulation. 2005 Aug 30;112(9 Suppl):I178-83. doi: 10.1161/CIRCULATIONAHA.104.522292. PMID 16159812
- [Background] Kawamoto A, Asahara T, Losordo DW. Transplantation of endothelial progenitor cells for therapeutic neovascularization. Cardiovasc Radiat Med. 2002 Jul-Dec;3(3-4):221-5. doi: 10.1016/s1522-1865(03)00082-9. PMID 12974378
- [Background] Kawamoto A, Tkebuchava T, Yamaguchi J, Nishimura H, Yoon YS, Milliken C, Uchida S, Masuo O, Iwaguro H, Ma H, Hanley A, Silver M, Kearney M, Losordo DW, Isner JM, Asahara T. Intramyocardial transplantation of autologous endothelial progenitor cells for therapeutic neovascularization of myocardial ischemia. Circulation. 2003 Jan 28;107(3):461-8. doi: 10.1161/01.cir.0000046450.89986.50. PMID 12551872
- [Background] Kawamoto A, Iwasaki H, Kusano K, Murayama T, Oyamada A, Silver M, Hulbert C, Gavin M, Hanley A, Ma H, Kearney M, Zak V, Asahara T, Losordo DW. CD34-positive cells exhibit increased potency and safety for therapeutic neovascularization after myocardial infarction compared with total mononuclear cells. Circulation. 2006 Nov 14;114(20):2163-9. doi: 10.1161/CIRCULATIONAHA.106.644518. Epub 2006 Oct 30. PMID 17075009
- [Background] Peichev M, Naiyer AJ, Pereira D, Zhu Z, Lane WJ, Williams M, Oz MC, Hicklin DJ, Witte L, Moore MA, Rafii S. Expression of VEGFR-2 and AC133 by circulating human CD34(+) cells identifies a population of functional endothelial precursors. Blood. 2000 Feb 1;95(3):952-8. PMID 10648408
- [Background] Ma N, Ladilov Y, Kaminski A, Piechaczek C, Choi YH, Li W, Steinhoff G, Stamm C. Umbilical cord blood cell transplantation for myocardial regeneration. Transplant Proc. 2006 Apr;38(3):771-3. doi: 10.1016/j.transproceed.2006.01.061. PMID 16647467
- [Background] Yin AH, Miraglia S, Zanjani ED, Almeida-Porada G, Ogawa M, Leary AG, Olweus J, Kearney J, Buck DW. AC133, a novel marker for human hematopoietic stem and progenitor cells. Blood. 1997 Dec 15;90(12):5002-12. PMID 9389720